CLINICAL TRIAL: NCT05288114
Title: A Pilot Study of the Signal Relief Patch for the Treatment of Musculoskeletal Pain
Brief Title: Signal Relief Patch in Musculoskeletal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Signal Relief (Industry)
Collaborators: Proxima CRO (Industry); ITC Imaging, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Signal -01-21
Record Dates: First submitted 2022-01-24; First posted 2022-03-18 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-01

CONDITIONS: Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Signal Relief Patch — Eligible subjects will be provided a Signal Relief patch, the instructions for use, and patch placement materials (adhesive, athletic tape, or wrap as applicable for the location of the pain). Subjects will be instructed to use the patch daily for seven days. The patch must be worn constantly except when showing or swimming.

SUMMARY:
assess the efficacy of the Signal Relief patch for the management of general musculoskeletal pain

DETAILED DESCRIPTION:
The Signal Relief Patch is an innovative, non-invasive technology that exists as a thin, flexible patch. The patch contains no drugs, wires, or batteries. Nano-capacitors utilized within the Signal Relief Patch were originally developed to replace military antenna systems with no additional power supply. Since development, it was incidentally found that these nano-capacitors may help control pain by working with the body's electrical system. Although the details of how these nano-capacitors facilitate the alleviation of pain are still under investigation, the possibility of reducing pain through a non-invasive, nonpharmacological method is extremely appealing.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject aged ≥ 18 years.
2. Currently seeking treatment for chronic musculoskeletal pain management.
3. Visual analog scale score > 4 at baseline.
4. Willing to refrain from the use of prescription pain medications during study participation.
5. Able and willing to provide informed consent.

Exclusion Criteria:

- 1. Receiving other investigational agents or on another clinical trial. 2. In emergent need for pain management. 3. Acute injury requiring rapid intervention or treatment. 4. The subject is using prescription medications (e.g., celecoxib, codeine, oxycodone, prednisone, etc.) for pain management regularly or PRN.

5. The subject is currently undergoing or planning to begin physical therapy. 6. The subject is planning to begin a new exercise routine. 7. Subject has implantable pain device, pacemaker, defibrillator, or other neuromodulation implantable device 8. Known to be pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-09-29 (Actual)

PRIMARY OUTCOMES:
% change in Pain Baseline to End | 7 days
  using visual analogue, proportion of subjects achieving at least a 30% reduction in reported pain on the visual analog scale score from baseline to the end of treatment.measurement and pain medication diary

SECONDARY OUTCOMES:
Improvement in brief pain inventory score baseline to end 0-10 scale; 0 being no pain, 10 being worst pain | 7 days
  proportional change in subject-reported scores on the Brief Pain Inventory Form
change in pain medication use baseline to end | 7 days
  subject-reported daily use of other medications intended for pain management using medication diary

OTHER OUTCOMES:
Exploratory | 7 days
  assess biomarker SubstanceP in response to study therapy

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Valley of the Sun Institute for Pain Management, Scottsdale, Arizona
  - Helios Health, Sedona, Arizona

IPD SHARING:
Plan to Share IPD: No